CLINICAL TRIAL: NCT03901209
Title: First-In-Man Performance and Safety Evaluation of the CARLO® Device in Midface Osteotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Osteotomy Tools (AOT) AG (Industry)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOT2019-01
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Abnormalities, Jaw; Malocclusion, Angle Class III
MeSH Terms: conditions — Jaw Abnormalities; Malocclusion, Angle Class III | interventions — Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: The study design is a prospective, bi-national, multi-center (3 centers), open-label single arm, confirmatory clinical study - with an initial explorative sequential phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laser osteotomy (Experimental): The planned mid-face osteotomy (e.g. LeFort I) is performed using the CARLO osteotomy device, where a patient-specific intervention plan based on preoperative imaging is loaded on the system to allow the device to show and suggest a location for the osteotomy.
  Interventions: Device: Mid-face osteotomy

INTERVENTIONS:
Device: Mid-face osteotomy — The mid-face osteotomy - typically according to LeFort I - is performed using a pulsed erbium-doped yttrium aluminium garnet (Er:YAG) laser driven by the CARLO robot arm.
  Other Names: Orthognathic Surgery, LeFort I

SUMMARY:
The study product is a Cold Ablation Robot-guided Laser Osteotome (CARLO®) robotic surgery device. It is a device that removes hard tissue such as bone by means laser ablation - it is therefore an alternative to Piezo-Electric osteotomes and/or oscillating saws or other mechanical instruments for bone cutting. In this study, the CARLO device is integrated with a computer-assisted pre-operative planning and intra-operative navigation, and will be used for Patients requiring an orthognathic procedure with a mid-face osteotomy, for whom a procedure plan is defined based on preoperative imaging.

DETAILED DESCRIPTION:
The objective of this first-in-man study is to confirm the performance and safety of the CARLO® robotic surgery device (manufactured by Advanced Osteotomy Tools SA) for the execution of preoperatively planned midface osteotomies.

The study is designed and powered to confirm, in clinical use across multiple sites, that the CARLO® device can be used to accurately perform straight-line mid-face osteotomies according to preoperative plans, and with results and a safety profile that are comparable to current state-of-the-art osteotomy methods. Multiple risk mitigations are in place to ensure safety, especially for the initially enrolled patients.

A postoperative follow-up of up to 28 days will be included in this study, in order to assess initial soft tissue healing and recovery, and to enable the identification of any soft-tissue injuries that would not have been immediately apparent.

After end of study of each individual patient, safety monitoring will go on for the duration of the study until the last visit of the last patient.

ELIGIBILITY:
Inclusion Criteria:

[ Indication for performing a mid-face osteotomy using a transoral approach, and suitability for use of CARLO® system: ]

1. Surgical relocation of the maxilla is indicated, using a mid-face osteotomy via a transoral approach that can be performed using bilateral straight-cut lines (LeFort I). Patients for whom a concomitant re-positioning of the mandibula or other corrections are indicated may be included in the study, as long as these corrections do not affect the repositioning of the maxilla that is being assessed; these additional osteotomies will not be performed using the CARLO® system.

   [ General requirements related to enrollment in a clinical study ]
2. Patient is willing and able to attend all scheduled visits and comply with all study procedures
3. Aged ≥18
4. Ability to understand and give study-specific informed consent
5. Written informed consent obtained from patient [ General precondition for orthognathic surgery ]
6. Proven completion of the facial growth

Exclusion Criteria:

[ General contraindications related to enrollment in a clinical study ]

1. Female patients who are pregnant or breast feeding or are planning to become pregnant during the study
2. Other patients who are vulnerable persons, such as adults lacking the capacity in the consent procedure, patients in emergency situations.
3. Known or suspected non-compliance, drug or uncontrolled alcohol abuse.
4. Presence of any condition or abnormality that in the opinion of the Investigator of the Investigator would compromise the safety of the patient or quality of the data
5. The patient is participating in, or intends to participate in another investigational drug or device clinical trial within 12 months after enrollment
6. Enrolment of the Investigator, his/her family members, employees and other dependent persons [ General contraindications for orthognathic surgery ]
7. Missing indication for orthognathic surgery
8. Patients with bleeding diathesis or coagulopathy
9. Patients with increased perioperative airway risk factors due to anatomical structures which limits usage of endotracheal intubation
10. Patients with intolerance or hypersensitivity to local anesthetics
11. Patients with consumptive/malignant primary disease (e.g. renal failure, hepatic dysfunction, severe heart failure, etc.) and a life expectancy of < 6 months
12. Patients that have an odontogenic osteomyelitis
13. Patients that have a diagnosed bone metabolism disorder e.g. Osteoporosis, Osteomalacia, Paget's disease, renal osteodystrophy, parathyroid disorders
14. Patients who have received or are receiving antiresorptive therapy (bisphosphonates).
15. Patient has previously undergone radiotherapy in the region of the intended osteotomy
16. Patients with impaired wound healing, for example due to Type II diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Technical Success of Device Use | Upon completion of the procedure
  Successful use of the device through all required steps: initial set-up and self-test, selection of each osteotomy path, previsualization of the path, completion of the osteotomies, and system shut down.
RMS error during registration of in-situ patient with pre-operative model | Intra-operative observation
  Point-pair matching performed to match preoperative imaging with the in-situ patient could be completed with a Root Mean Square error that does not exceed 1.5 mm.
Position of the performed osteotomies is within 2 mm of the preoperatively planned location. | Intra-operative observation
  The postion of the performed osteotomies is measured intraoperatively, relative to (orthogonally located) landmarks selected on the preoperative 3D model. The oucome is successful if this distance does not exceed 2 mm.
Successful completion of the maxillary downfracture and procedure without unusual difficulties. | Intra-operative observation
  The maxillary mobilization (pterygo-maxillary disjunction, pull-down fracture) can be completed as usual. No difficulty is encountered that is unusual for the procedure.

SECONDARY OUTCOMES:
Key variables of the osteotomy procedures (durations) | Upon completion of the procedure
  Variables assessed include:
  1. Duration of overall osteotomy procedure (first skin incision to skin closure).
  2. Duration of patient registration with the CARLO® device (from on-screen selection of first point to be matched to display of an accepted Root Mean Square Error value).
  3. Duration of CARLO® device cutting for each osteotomy.
Absence of unusual complications that delay initial patient discharge. | 1 week post-procedure
  Overall well-being of the patient allows a normal discharge from the hospital without unusual delay (within one week).
Absence of unusual soft tissue healing difficulties (14 days status). | 2 weeks post-procedure
  During the visit scheduled at 14 days, soft tissue healing allows the removal of stitches as normally possible.
Absence of healing anomalies during final visit (28 days status) | 4 weeks post-procedure
  During the visit scheduled at 28 days, absence of any anomaly or concern related to post-operative healing.
Accuracy of the execution of the planned osteotomy based on postoperative imaging | Assessed ~2 weeks postoperatively based on postoperative imaging (CBCT)
  Accuracy of the performed cut measured on postoperative CT (distance of the cut start and end relative to the incisor point and to the ipsilateral mesio-buccal cuspid, respectively). Target is to perform cut within 2 mm of the planned position.
Accuracy of the final maxilla location, compared to plan, based on postoperative imaging | Assessed ~2 weeks postoperatively based on postoperative imaging (CBCT)
  Accuracy of the maxilla relocation, comparing on CT imaging the position of five defined landmarks (e.g. incisor point, tips of the upper canines, tips of the mesio-buccal cuspid) between the plan and the final result.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Müller, Principal Investigator — Universitätsspital Basel; Marcello Augello, Principal Investigator — Kantonsspital Aarau
Locations (4):
- Allgemeines Krankenhaus der Stadt Wien (AKH Wien), Vienna, Austria
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Switzerland (2):
  - Kantonsspital Aarau AG, Aarau, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City

IPD SHARING:
Plan to Share IPD: No